CLINICAL TRIAL: NCT01254877
Title: Ondansetron Pharmacotherapy for Hazardous Drinking in HIV+, African-American Women
Brief Title: Ondansetron, Alcohol Use, and Alcohol-Related Symptoms In HIV+ Persons
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NA_00032774; R01AA018896 (NIH)
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Results first posted 2018-04-17 (Actual); Last update posted 2018-04-17 (Actual); Status verified 2018-03

CONDITIONS: Alcohol Abuse; Alcohol Dependence
Keywords: HIV
MeSH Terms: conditions — Alcoholism | interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Ondansetron - sugar pill (Placebo Comparator): Placebo is an oral preparation made to appear and taste like the active drug preparation.
  Interventions: Drug: placebo ondansetron
- low dose ondansetron (0.2 mg bid) (Experimental)
  Interventions: Drug: ondansetron
- moderate dose ondansetron (0.8 mg bid) (Experimental)
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: ondansetron — ondansetron 0.2 mg bid, oral preparation, 16 weeks
  Arms: low dose ondansetron (0.2 mg bid)
Drug: placebo ondansetron — Matching placebo will be prepared using a colorless strawberry syrup, simple syrup and flat Schweppes tonic water.
  Arms: Placebo Ondansetron - sugar pill
Drug: Ondansetron — Ondansetron 0.8 mg bid, oral preparation, 16 weeks duration
  Arms: moderate dose ondansetron (0.8 mg bid)

SUMMARY:
The proposed randomized clinical trial will investigate a novel pharmacotherapy for hazardous drinking, HIV-infected men and women, using the serotonin receptor (5-HT3) antagonist ondansetron. The investigators predict that participants who are treated with active doses of ondansetron will reduce their drinking more and show better HIV treatment participation and progress compared to participants who are treated with placebo. This study will provide important new safety and efficacy results on drinking and HIV outcomes following alcohol pharmacotherapy in HIV-infected persons.

DETAILED DESCRIPTION:
Hazardous drinking is particularly harmful in HIV-infected persons. It impairs the immune system, accelerates HIV disease progression, slows initiation of antiretroviral therapy (ART) and decreases adherence. Thus, the development of effective alcohol treatments for this clinical population is particularly important. The investigators are proposing to investigate the effectiveness of ondansetron pharmacotherapy for the treatment of hazardous alcohol use and alcohol abuse/dependence among HIV-infected patients. Ondansetron, a 5-HT3 antagonist, will be studied for several reasons: 1) evidence of effectiveness in persons who want to cut-down or reduce their drinking and who are not abstinent at medication initiation; 2) moderate-to-strong effects among early onset problem drinkers, a characteristic that is over represented in our clinic patients; 3) a very mild side-effect profile, making it an ideal pharmacotherapy candidate in patients who are often receiving multiple other medications with significant side-effects; and 4) its primary indication is for treatment of nausea, a common side-effect of antiretroviral (ARV) medications.

The proposed study is a placebo-controlled, randomized clinical trial of ondansetron for the treatment of hazardous drinking and alcohol use disorders among HIV-infected patients recruited from the Baltimore/Washington area. Participants will be genotyped for a functional polymorphism of the serotonin transporter gene. They will be randomized to one of three treatment groups: placebo, low dose ondansetron (0.2 mg bid) and moderate dose ondansetron (0.8 mg bid). All subjects will undergo 16 weeks of pharmacotherapy in combination with medication management, and will be followed for 3 and 6 months after medication has ended.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be at least 18 years old and HIV-infected
* All subjects will be actively drinking at hazardous levels (1) AUDIT score => 4 for women or =>8 for men, or 2) => 2 binge drinking episodes/month, or 3) >7 drinks/week for women or >14 drinks/week for men)

Exclusion Criteria:

* Liver Function Tests (LFTs) > 5 X normal
* Magnesium or potassium > 3 X normal
* Qtc => .460 and or a family history of long QT syndrome (LQT)
* Inability to read and comprehend English
* Actively psychotic or other severe mental health symptoms that would prevent appropriate participation
* Current enrollment in alcoholism treatment program
* Pregnancy; Ondansetron is currently a category B drug. While animal data have not identified any harmful effects to mother or fetus, there have not been adequate human controlled trials to recommend routine use in this population

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 357 (Actual)
Dates: Start 2010-12; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E McCaul, Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Johnson BA, Roache JD, Javors MA, DiClemente CC, Cloninger CR, Prihoda TJ, Bordnick PS, Ait-Daoud N, Hensler J. Ondansetron for reduction of drinking among biologically predisposed alcoholic patients: A randomized controlled trial. JAMA. 2000 Aug 23-30;284(8):963-71. doi: 10.1001/jama.284.8.963. PMID 10944641

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 357 persons signed informed consent; 205 were randomized. 137 exclusions were mainly due to insufficient alcohol use (as determined by self-report or biomarker), abnormal QT interval, or significant mental health symptoms that precluded assessment completion. An additional 13 participants withdrew, were discontinued by the investigators or died.
Period: Overall Study
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
Started | 67 | 69 | 69
Completed | 57 | 58 | 64
Not Completed | 10 | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid) | Total
Number analyzed (Participants) | 67 | 69 | 69 | 205
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.7 (8.7) | 48.7 (8.2) | 47.8 (9.5) | 48.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 23 | 27 | 71
  Male | 46 | 46 | 42 | 134
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 65 | 66 | 64 | 195
  Other | 2 | 3 | 5 | 10
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 69 | 69 | 205
Number of drinks per drinking day [Mean (Standard Deviation); unit: standard alcohol drink] | 9.1 (5.5) | 10.5 (7.7) | 10.0 (8.7) | 9.9 (7.3)
Number of days abstinent from alcohol/week [Mean (Standard Deviation); unit: days/week] | 2.9 (1.9) | 3.0 (2.1) | 3.3 (1.9) | 3.1 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: Number of Alcoholic Containing Drinks Per Drinking Day
Description: The Time-line Follow-back (TLFB; Sobell, Sobell, Leo & Cancilla, 1988) is conducted as an interview administered by trained and certified research staff. The interview obtains participant self-reports of daily drinking, including number and type of alcoholic beverages. These data are used to quantify an individual's drinking pattern including the number of drinks per drinking day and drinking frequency. The TLFB was completed biweekly and quantified over the 16-week medication period
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: Standard alcohol drinks per drinking day
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
Number analyzed (Participants) | 67 | 69 | 69
Standard alcohol drinks per drinking day | 5.9 (3.8) | 6.1 (4.3) | 5.9 (3.9)

2. Primary Outcome: Number of Days/Week Abstinent From Alcohol
Description: The Time-line Follow-back (Sobell, Sobell, Leo & Cancilla, 1988) is used to obtain this secondary dependent measure. Alcohol use will be assessed biweekly and quantified over the 16-week medication period. Number of days/week abstinent from alcohol is calculated as the number of abstinent days divided by the number of study medication days (adjusted for days in confinement (e.g., hospitalization; jail)) and multiplied by 7.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: days/week abstinent from alcohol
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
Number analyzed (Participants) | 67 | 69 | 69
days/week abstinent from alcohol | 4.7 (2.2) | 4.9 (2.0) | 4.8 (2.2)

3. Secondary Outcome: Medication Safety
Description: Medication side-effects and adverse events were measured using the Systematic Assessment for Treatment of Emergent Events (SAFTEE). The SAFTEE contains 25 detailed questions that systematically address 29 body systems. A trained interviewer elicits information about onset, duration, pattern, and judgment of attribution. For the present trial outcome, we report number of events.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: number of events
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
Number analyzed (Participants) | 67 | 69 | 69
number of events | 11.4 (11.1) | 12.4 (13.4) | 11.0 (12.3)

4. Secondary Outcome: Number of Subjects Who Discontinue Due to Side Effects
Description: The investigators will count the number of subjects who discontinue medication during the 16-week intervention period due to complaints of side effects.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
Number analyzed (Participants) | 67 | 69 | 69
Participants | 0 | 0 | 0

5. Secondary Outcome: Alcohol-related Problems
Description: Alcohol-related problems were measured using the Short Inventory of Problems - revised (SIP-R), a self-report inventory of adverse consequences associated with alcohol and drug use. The SIP instructs participants to indicate how often each of 15 consequences has occurred during the past three months ("never," "once or a few times," "once or twice a week," "daily or almost daily"; scored 0-3). Item responses are summed to produce a total score and five subscale scores. Total scores range from 0 - 45.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
Number analyzed (Participants) | 67 | 69 | 69
units on a scale | 6.6 (7.3) | 7.5 (7.9) | 8.3 (15.7)

6. Secondary Outcome: HIV Medication Adherence
Description: The investigators will obtain patient self reports of the number of HIV medication doses taken as a function of the total number of doses prescribed. The adherence measure is expressed as the % of prescribed doses.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: percentage of prescribed doses
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
Number analyzed (Participants) | 67 | 69 | 69
percentage of prescribed doses | 92.4 (31.6) | 87.6 (37.6) | 85.4 (31.7)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo Ondansetron - Sugar Pill | Low Dose Ondansetron (0.2 mg Bid) | Moderate Dose Ondansetron (0.8 mg Bid)
All-Cause Mortality (participants affected / at risk) | 1/67 | 0/67 | 1/69
Serious Adverse Events (participants affected / at risk) | 16/67 | 20/69 | 5/69
Other Adverse Events (participants affected / at risk) | 7/67 | 5/69 | 8/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Ondansetron - Sugar Pill (N=67) | Low Dose Ondansetron (0.2 mg Bid) (N=69) | Moderate Dose Ondansetron (0.8 mg Bid) (N=69)
Acute Alcohol Intoxication (Psychiatric disorders) | 2 (2) | 6 (6) | 0 (0) — Acute alcohol intoxication treated in the Emergency Dept or inpatient hospitalization
Pneumonia/Respiratory Infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (5) | 1 (1)
Psychiatric disorder (Psychiatric disorders) | 2 (2) | 2 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2) | 0 (0)
cardiovascular event (Cardiac disorders) | 4 (4) | 1 (1) | 0 (0)
Other (General disorders) | 2 (2) | 5 (5) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Ondansetron - Sugar Pill (N=67) | Low Dose Ondansetron (0.2 mg Bid) (N=69) | Moderate Dose Ondansetron (0.8 mg Bid) (N=69)
Cough/cold symptoms (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 4 (4)
Alcohol intoxication/withdrawal (Psychiatric disorders) | 2 (2) | 1 (1) | 1 (1)
Rash/wound infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Other (General disorders) | 1 (1) | 2 (2) | 1 (1)

LIMITATIONS AND CAVEATS:
Drinking data are based on patient self-report.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No